CLINICAL TRIAL: NCT00527657
Title: A Phase I Study of Temozolomide, Thalidomide, and Lomustine (TTL) in Patients With Metastatic Melanoma in the Brain
Brief Title: Temozolomide, Thalidomide, and Lomustine (TTL) in Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0595; NCI-2012-01587 (Registry Identifier: NCI CTRP); NCT01867619 (obsolete NCT alias)
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Brain Neoplasms; Melanoma
Keywords: Brain Neoplasms; Melanoma; Metastatic Melanoma; Brain Metastasis; Temozolomide; Temodar; Thalidomide; Thalomid; Lomustine; CCNU; CeeNU
MeSH Terms: conditions — Brain Neoplasms; Melanoma | interventions — Lomustine; Temozolomide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lomustine + Temozolomide + Thalidomide (Experimental): Lomustine starting dose 30 mg/m^2 by mouth daily on Day 1 and 29. Temozolomide 75 mg/m^2 by mouth daily on Days 1 to 42. Thalidomide 200 mg/m^2 by mouth daily.
  Interventions: Drug: Lomustine; Drug: Temozolomide; Drug: Thalidomide

INTERVENTIONS:
Drug: Lomustine — Starting dose 30 mg/m^2 by mouth daily on Day 1 and 29.
  Other Names: CCNU; CeeNU
Drug: Temozolomide — 75 mg/m^2 by mouth daily on Days 1 to 42.
  Other Names: Temodar
Drug: Thalidomide — 200 mg/m^2 by mouth daily.
  Other Names: Thalomid

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of lomustine (CCNU, CeeNUTM) that can be given with temozolomide (TemodarTM) and thalidomide (ThalomidTM) in the treatment of metastatic melanoma that has spread to the brain. The safety and effectiveness of this combination therapy will also be studied.

DETAILED DESCRIPTION:
Temozolomide works by blocking a tumor cell's ability to grow. Lomustine is also a chemotherapy drug that works by killing tumor cells. Studies have shown that when lomustine and temozolomide are given together, they decrease the amount of a certain protein, allowing the tumor cells to be more easily killed. Thalidomide is a drug that alters the immune system. it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

If you are found to be eligible to take part in this study, you will begin treatment. All 3 drugs will be taken by mouth at home. Each treatment cycle will last for 8 weeks. You will take temozolomide once a day for 6 weeks followed by two weeks off. The best time to take temozolomide is around bedtime, since you must not eat for at least 1 hour before and 1 hour after taking it. The number of capsules you will take is based on your height and weight. You must swallow all the temozolomide capsules at the same time with 8 ounces of water (do not chew them).

You will take thalidomide every day for the entire 8-week cycle. Thalidomide should also be taken near bedtime, usually 30 to 45 minutes before the temozolomide dose. If you are under 70 years of age, you will start at a set dose and take the same dose throughout the study. If you are age 70 or over, the dose will start lower and will increase every 2 weeks until you are taking the prearranged set dose that those under the age of 70 are taking. Your doctor will be watching for side effects as the dose increases and may keep you at a lower dose if necessary.

In the first groups of patients (3-6 patients per group, total up to 18 patients) to be enrolled, each new group of participants will be given a higher dose of lomustine than the previous group until the highest safe dose of lomustine is found or until 18 patients have been enrolled. Responses to these doses will be evaluated. Once the best dose is found, all future participants will receive that dose of lomustine.

You will take 2 doses of lomustine every 8 weeks. You will take the first dose of lomustine on Day 1 of the 8-week cycle. You will take the second dose, which will be half as big as the first dose, on Day 29 (the day after the first 4 weeks) of the 8-week cycle. The dose of lomustine is also based on your height and weight. Lomustine should be swallowed and not chewed.

During treatment, every 2-4 weeks, you will have a complete physical exam and blood drawn for testing (1-2 tablespoons). These tests will let the doctor know if the treatment should be changed, briefly interrupted, or stopped. Women who are able to have children must have a negative pregnancy test every week for the first 4 weeks if they have regular menstruation and every 2 weeks if their periods are irregular.

At the end of 8 weeks, you will have x-rays or scans done again to see how the tumors have responded. If they are the same size or have gotten smaller, you may continue the treatment. You may stay on treatment as long as you are not having severe side effects and your tumor is either staying the same size or getting smaller. Treatment will be stopped if the tumors are getting bigger.

If you are withdrawn from the study for any reason you will be contacted by phone every three months to learn how are you doing health wise.

This is an investigational study. None of the 3 drugs used in this study have been approved by the FDA for the treatment of melanoma. Temozolomide has been approved for the treatment of brain cancer. Thalidomide has not yet been approved for the treatment of cancer. Lomustine is approved for the treatment of brain tumors and Hodgkin's disease. All of the drugs are commercially available. Their use together in this study is experimental.

Up to 18 patients will take part in this Phase I portion of the study, and another 30 patients in Phase II if progresses, with up to 48 patients total. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic Documentation: Histologic or cytologic diagnosis of distant metastatic melanoma and clinical evidence of brain metastasis.
2. Pts must have brain lesions of =/> 1.0cm longest dimension by MRI or spiral CT, if MRI not feasible or > 0.5cm by MRI with 3D images. Pts with/without extracranial disease are eligible. Measurable extracranial disease is not required. Lesions that are considered non-measurable include: <1.0 cm by MRI or Spiral CT, Bone lesions, Leptomeningeal disease, Ascites, Pleural/pericardial effusion, Lymphangitis cutis/pulmonis, Abdominal masses that are not confirmed and followed by imaging techniques, Cystic lesions, lesions that are in a previously irradiated area, unless new growth can be documented.
3. Age >/= 18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status: 0 or 1
5. No more than 1 prior chemotherapy regimen and no prior chemotherapy for brain metastases. No prior treatment with continuous daily dose of temozolomide; prior immunotherapy and surgical resection are permitted. Patients with prior history of whole brain radiotherapy (WBRT) and stereotactic radiosurgery (SRS) are permitted providing that there is measurable lesion with documented growth post radiation or new disease.
6. (#5 continued) Progression of lesions treated with WBRT must be shown by 2 post treatment brain imaging at least 3 weeks apart. Progression of disease is also considered when the patient had increase of lesions as per MRI of brain obtained 4 weeks or more after WBRT completed when compared to baseline MRI obtained less than 1 week prior to start of radiation. Lesions treated with SRS must have responded and then progressed.
7. The following time periods must have elapsed since prior therapy: 3 weeks since surgical resection or stereotactic radiosurgery; 4weeks since prior whole brain radiation therapy; 6 weeks since prior nitrosureas or mitomycin C. Biologic agents used as adjuvants and vaccines or cellular therapies will not require 4-week wash out period if the patient meets all eligibility criteria.
8. No frequent vomiting and/or medical condition that could interfere with oral medication intake (e.g., partial bowel obstruction).
9. No other concurrent chemotherapy/immunotherapy/radiotherapy.
10. No history of active angina or myocardial infarction within 6 months. No history of significant ventricular arrythmia or uncontrolled arrythmia or bradycardia. The study participants must have resting heart rate of 48 or greater (.e.i - to receive Thalidomide).
11. No prior history of deep vein thrombosis (DVT) or pulmonary embolism (PE).
12. No known HIV disease. Patients with a history of intravenous drug abuse or any other behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus. Because peripheral neuropathies are a common toxicity of antiviral therapy and of viral infection in HIV patients, as well as a common significant toxicity with thalidomide, patients who test positive or who are known to be infected are not eligible. An HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk.
13. No pre-existing neuropathy that is >/= grade 2, including uncontrolled seizures.
14. No expected need for radiotherapy to brain or any extracranial metastatic site during the period of participation in the study.
15. Patients may not be taking Coumadin, warfarin or heparin products or their derivatives.
16. Patients who require anti-platelet therapy such as daily aspirin, Plavix or ibuprofen are not eligible to participate.
17. Patients requiring the use of bisphosphonates (e.g., zoledronic acid) are not eligible to participate. Patients who receive thalidomide in combination with zoledronic acid are potentially at increased risk of renal dysfunction.
18. Required Initial Laboratory Data: Granulocytes >/= 1,500/ml; Platelet count >/= 100,000/ul; Creatinine </=2 mg/dl; Transaminases (ALT,AST) </= 3 * upper limits of normal; Alkaline phosphatase </= 3 * upper limits of normal; thyroid-stimulating hormone (TSH) Within normal limits Serum beta-HCG Negative (in female patients unless S/P hysterectomy or menopausal or no menses for 24 months). Assay must have a sensitivity of at least 50 mIU/ml. Serum anticonvulsant levels (for patients on a measurable anticonvulsant) must be within therapeutic range. EKG must be without acute abnormalities or uncontrolled arrhythmia.
19. Pregnant and nursing women are not eligible for treatment on this protocol. Women of childbearing potential must agree to abstain from all intercourse or use two methods of birth control for 28 days prior to treatment and while under treatment with thalidomide and for 4 weeks after completing therapy. One of the methods of birth control must be highly active (IUD, hormonal, tubal ligation or partner's vasectomy) and used concomitantly with one additional method(e.g., latex condom, diaphragm or cervical cap. Please see also eligibility criteria 19 and 20.
20. In addition, women of childbearing potential must have morning urine b-HCG performed within 1 week prior to registration and within 24 hours before beginning study treatment. All the precautions for childbearing potential women are required even in patients with infertility unless due to hysterectomy or the patient has been post menopausal (has had no menses for at least 24 consecutive months). Men must agree to abstain from unprotected sexual intercourse. Male patients should request that female partners use a second method of birth control in addition to the male barrier method (condoms).
21. All patients (men and women) must agree to use medically approved contraceptive measures simultaneously prior to starting thalidomide therapy, all during drug therapy, and for at least 1 month after therapy has stopped. Women of childbearing potential should start using medically approved contraceptive measures 4 weeks prior to starting thalidomide therapy.
22. Patients must give written consent.
23. Patients must be willing and able to comply with the FDA-mandated S.T.E.P.S version 3 program.

Exclusion Criteria:

1. Presence of any ongoing toxic effect from prior treatment.
2. Serious infection requiring intravenous antibiotics, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
3. Concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies, but which have not required anti-tumor treatment within the preceding 24 months will be allowed to enter the trial. Patients with a history of a T1a or b prostate cancer (detected incidentally at transurethral prostatectomy (TURP) and comprising less than 5% of resected tissue) may participate if the prostate-specific antigen (PSA) remained within normal limits since TURP.
4. Any other medical condition or reason that, in the principal investigator's opinion, makes the patient unsuitable to participate in a clinical trial including but not limited to active bleeding, prior surgical procedures affecting absorption or gastrointestinal tract disease resulting in inability to take oral medication.
5. Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-02-09; Primary Completion 2012-02-02 (Actual); Study Completion 2012-02-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 1 cycle (8 weeks) of therapy

SECONDARY OUTCOMES:
Objective (CR+PR) response rate at the MTD | 1 cycle (8 weeks) of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E. Papadopoulos, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Web Site — http://www.mdanderson.org